CLINICAL TRIAL: NCT07364097
Title: Does Eliminating Alarm Noise Cacophony for Intensive Care Staff and Patients Improve Burnout and Encephalopathy Levels
Brief Title: A Study of Silent Alarm Delivery Versus Standard Audible Alarm Delivery in Intensive Care and High Dependency Units
Acronym: DECIBEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MindWave Medical Inc (Industry)
Responsible Party: Principal Investigator, Daniel F Niendorff, MD, MindWave Medical Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: D26
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Delirium in the Intensive Care Unit; Burnout, Healthcare Workers; Noise in the ICU; Alarm Fatigue; Alarm Fatigue in Intensive Care Unit Nurses; Alarms; Nursing Workload
Keywords: ICU delirium; alarm fatigue; silent alarm; alarm noise; nursing burnout; nursing work; alarm response
MeSH Terms: conditions — Burnout, Psychological; Alert Fatigue, Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silent alarm strategy (Experimental): The intervention consists of the implementation of a silent alarm system for the clinical environment. The silent alarm system consists of a self-locating interface device, which is interposed between an alarm-generating device and its audio output. This device contains communication, locating, motion, logic, and relay chips, which enable the interface device to identify its location and staff responsible for that location, as well as to detect audio output from the alarm-generating device, and to control the audible state of that output. The Interface device can communicate with separate bone conduction headsets worn by staff, which contain sensors that confirm staff presence at the headset, and buttons for response to an alarm announcement. The interface device then delivers alarms silently to those staff specifically responsible for its location when a responsible staff member can be identified, confirmed to be present, and accepts responsibility for the alarm through button action
  Interventions: Other: Silent alarm strategy
- Control (No Intervention): In the control arm of the study, interface devices (as described in the experimental arm) will remain in place for data collection only, but will allow all alarms to be audible, and will not attempt silent alarms.

INTERVENTIONS:
Other: Silent alarm strategy — The intervention consists of the implementation of a silent alarm system in the clinical environment. The silent alarm system consists of a self-locating interface device, which is interposed between an alarm-generating device and its audio output. This device contains communication, locating, motion, logic, and relay chips, which enable the interface device to identify its location and staff responsible for that location, as well as to detect audio output from the alarm-generating device, and to control the audible state of that output. The Interface device can communicate with separate bone conduction headsets worn by staff, which contain sensors that confirm staff presence at the headset, and buttons for response to an alarm announcement. The interface device then delivers alarms silently to those staff specifically responsible for its location when a responsible staff member can be identified, confirmed to be present, and accepts responsibility for the alarm through button action.
  Arms: Silent alarm strategy

SUMMARY:
The goal of the trial is to learn if a strategy to eliminate audible alarm noise in intensive care and high dependency units can reduce overall noise levels, patient delirium, staff alarm fatigue, and staff burnout. Researchers will implement a silent alarm strategy in specific care units for four weeks and compare this to a separate 4 weeks where a silent strategy is not implemented. Noise, burnout, delirium levels, and staff alarm response times will be compared between the silent and non-silent units.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Intensive or high dependency care unit.

Exclusion Criteria:

* Pre-existing diagnosis of dementia
* Endotracheally intubated (may enroll when extubated)
* CNS injury, infection, or malignancy as reason for admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Confusion Assessment Method - (CAM-S long form) | The CAM-S long form will be recorded every 12 hours during the four-week experimental period and also every 12 hours during the four-week control period.
  The CAM-S Long form is a structured assessment to evaluate the presence and severity of delirium. It consists of a structured clinical assessment that has proven to be reproducible and an accurate measure of delirium presence and severity. The CAM-S has a scoring range of 0-19 with higher scores indicating a greater severity of delirium.
Unit noise levels (Decibels) | 10 seconds Decibel measurement periods will be recorded consecutively for two four-week periods, consisting of the four-week intervention period, and the four-week control period.
  Unit noise levels will be recorded using an integrating Decibel monitor measuring 10 second periods for A-weighted equivalent sound pressure levels (LA-EQ), and also C-weighted peak sound pressure (LC-Peak) for those same 10 second periods. Both LA-EQ and LC-Peak will be averaged, and reported on the Decibel scale, a logarithmic scale of sound pressure levels from 0 Db(least sound pressure) to 194 Db (maximum measurable sound pressure).
Alarm Fatigue | The staff response times will be measured (in seconds) for every alarm occurring during the four-week intervention and control periods.
  Alarm fatigue is an involuntary learned response among staff alarm responders that occurs over time. When presented with a high frequency of alarms which either lack specificity of the condition to which they intend to call attention, or which have a low frequency of required staff intervention ("nuisance alarms"), staff response times become extended, and in some cases, responses do not occur at all. This trial will track staff response time as the time from alarm initiation to staff button response, or alarm audio termination.
  Alarm fatigue, assessed as the response time from alarm initiation to staff response (headset button response) or alarm audio termination, measured in seconds on every alarm occurring on every participating device during the study and control periods, each lasting four weeks. Time points for recording responses will be determined by alarm occurrence. Response times for the study and control periods will be averaged and compared statistically.

SECONDARY OUTCOMES:
Nursing Work | Two four-week periods consisting of one four-week period as active intervention unit, and one four-week period as control unit.
  Nursing Work - Pedometer Measurements. All nurses in each participating unit will wear a pedometer during work shifts. Pedometers will record the number of steps taken during each shift. At the end of each shift, nurses will record the number of steps taken, and the length of the shift (hours). At the end of each four-week period as either study or control, the total number of steps recorded for nursing shifts in that unit will be divided by the total number of shift hours recorded in that unit over the four-week period, to determine the average hourly step count for that unit during the four-week period of either study or control unit.
Total Audio Time | Two four-week periods consisting of one four-week period for each unit as control arm, and one four-week period for each unit as intervention arm.
  The time that audio equipment generates an audio signal will be monitored and recorded. The total cumulative duration (in hours, minutes and seconds) that all monitored medical equipment generates audio output signals in the observed unit will be recorded for two four-week periods consisting of one four-week period while the unit serves as control, and a separate four-week intervention period.
Use of medications intended to treat agitation | Cumulative doses of haloperidol and dexmedetomidine administered to all participants up to day 28 of the intervention and control periods.
  Use of haloperidol or dexmedetomidine
Artificial intelligence observed rest | Artificial intelligence observed rest will be monitored every 10 minutes for two four-week periods, consisting of the four-week control period and the four-week intervention period.
  A camera based artificial intelligence system will observe sleep/wake appearance every 10 minutes in both intervention and control units for the two four-week study periods. This system has been trained to observe and differentiate the appearance of sleep and wake. The system will track sleep and wake appearance for each individual every 10 minutes for the two complete four-week periods of study and intervention arms.

OTHER OUTCOMES:
Silent vs Audible alarm time | This proportional measurement will serve as a baseline for future investigators
  The total and proportional alarm time that equipment spent in audible and silent states will be recorded during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Niendorff, MD, Principal Investigator — MindWave Medical
Locations (1):
- Udayananda Multispecialty Hospital, Nandyāl, Andrah Pradesh, India

IPD SHARING:
Plan to Share IPD: No